CLINICAL TRIAL: NCT03852849
Title: Cohort Study on Appropriate Strategies of The Rapid Build of HIV Related Protective Barriers in Yunnan, China
Brief Title: Rapid Build of HIV Related Protective Barriers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Collaborators: Yunnan Center for Disease Control and Prevention (Other); Yunnan AIDS Care Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018ZX10721102-002
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Viral Suppression of HIV Infection
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- routine care group (No Intervention): Medical institutions will provide patients routine care according to the national program standard.
- medicine intervention group (Experimental): The dosage of 400 mg EFV will be used in the antiviral therapy.
  Interventions: Drug: The dosage of 400mg EFV
- consolidated intervention group (Experimental): Medical institutions will provide personal involved intervention strategies as well as the providing of dosage form of 400 mgEFV in their antiviral therapy.
  Interventions: Behavioral: Personal involved intervention strategies; Drug: The dosage of 400mg EFV

INTERVENTIONS:
Behavioral: Personal involved intervention strategies — Medical institutions will provide personal involved intervention strategies for patients which guided by viral load testing monthly until viral load drop below the detection limit.
  Arms: consolidated intervention group
Drug: The dosage of 400mg EFV — The dosage of 400mg EFV will be used in the antiviral therapy.
  Arms: consolidated intervention group; medicine intervention group

SUMMARY:
The purpose of the study is to screen the optimal intervention strategies to rapid establish the protective barriers against HIV-infection by maximally decreasing the viremia among HIV- infected patients.

DETAILED DESCRIPTION:
Sexual transmission became the primary route of HIV transmission in China and heterosexual transmission also contributed greatly to HIV epidemic which was mostly reported in South-west rural areas. In past years, Yunnan has experienced powerful campaign of scaling-up the HIV identification as well as antrertroviral therapy.

This study will investigate how to reach the last two of HIV'90-90-90 targets': to provide antiretroviral therapy (ART) for 90% of who diagnosed HIV infection and to achieve viral suppression for 90% of those treated.

The study population consists of participants who received an newly diagnosed HIV infection within the study period. All rerolled participants will be randomized into different study group. In intervention group, medical institutions will provide patients personal involved intervention strategies which guided by frequent viral load detection, and providing of the dosage form of 400 mg EFV in their antiviral therapy.

Main assessment measures are viral suppression rate of HIV-infected patients and treatment coverage .

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive participants who received an newly diagnosed HIV infection within the study period
* Having a current residential address inside of pilot site limits
* Eighteen years old or above
* HIV transmission is heterosexual contact

Exclusion Criteria:

* IDU
* Having severe mental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Viral suppression of HIV-infected patients | 12 months

SECONDARY OUTCOMES:
Treatment coverage | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Yan, PHD, Principal Investigator — National Center for AIDS/STD Control and Prevention
Locations (2):
- China (2):
  - Lincang Center for Disease Control and Prevention, Lincang, Yunnan
  - Wenshan Center for Disease Control and Prevention, Wenshan, Yunnan